CLINICAL TRIAL: NCT01041833
Title: Randomized Phase III Trial: Effect of All-trans Retinoic Acid With Chemotherapy Based on Paclitaxel and Cisplatin As First-line Treatment of Patients With Advanced Non-small Cell Lung Cancer and Expression of RAR-alfa and RAR-beta as Response Biomarkers
Brief Title: Effect of All-trans Retinoic Acid With Chemotherapy Based on Paclitaxel and Cisplatin As First-line Treatment of Patients With Advanced Non-small Cell Lung Cancer and Expression of RAR-alfa and RAR-beta as Response Biomarker
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Institute of Cancerología (Other Government)
Responsible Party: Oscar Arrieta, M.D., Department of Medical Oncology, Instituto Nacional de Cancerología
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CA/141/CB/563/09
Record Dates: First submitted 2009-09-07; First posted 2010-01-01 (Estimated); Last update posted 2010-01-01 (Estimated); Status verified 2009-09

CONDITIONS: Non Small Cell Lung Cancer
Keywords: All-trans retinoic acid; non-small cell lung cancer; retinoic acid receptor beta
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- atRA group (Experimental): atRA group will receive six cycles of 80 mg/m2 of cisplatin and 175 mg/m2 of paclitaxel plus atRA 45 m2/day before one week before treatment and during all the treatment
  Interventions: Drug: atRA
- Placebo Group (Placebo Comparator): Placebo group will receive six cycles of 80 mg/m2 of cisplatin and 175 mg/m2 of paclitaxel plus placebo before one week before treatment and during all the treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: atRA — atRA group will receive six cycles of 80 mg/m2 of cisplatin and 175 mg/m2 of paclitaxel plus atRA 45 m2/day before one week before treatment and during all the treatment
  Arms: atRA group
Drug: Placebo — Placebo group will receive six cycles of 80 mg/m2 of cisplatin and 175 mg/m2 of paclitaxel plus placebo before one week before treatment and during all the treatment
  Arms: Placebo Group

SUMMARY:
BACKGROUND Platinum-based chemotherapy (CT) is the standard treatment for advanced non-small-cell lung cancer (NSCLC). Unfortunately, the survival and response rate (RR) to CT is poor. There is great interest in new treatment strategies. One of this new strategies include the use of retinoids such as atRA. The synergistic effect of cytotoxic agents with retinoids has been demonstrated in lung cancer. At the INCan, our work group carried out a phase II study trial that included 107 patients with advanced NSCLC. They were randomized to receive atRA (20-mg/m2) or placebo combined with 80 mg/m2 of cisplatin and 175 mg/m2 of paclitaxel. The results showed a significant increase in the RR of the atRA group, reaching 55.8% ( 95% CI; 46.6-64.9%) compared with 25.4% (95% CI, 21.3-29.5%; p = 0.001) in patients who received placebo. Median Progression-free survival (PFS) in the atRA group was 8.9 months, while for those of placebo, PFS was 6.0 months (p = 0.008). There were no significant differences in the grade 3-4 side effects between groups, except for hypertriglycemia, which presented with greater frequency in the atRA group (p = 0.05). Immunohistochemical stains determine the RAR B2 expression in 6 of 60 tumor samples analyzed; however, all samples expressed RAR B2 in adjacent normal tissue.

HYPOTHESIS Patients with NSCLC who receive the scheme combined with first-line CT plus 45 mg/m2 of atRA will have a greater PFS and RR to CT with an acceptable toxicological profile.

OBJECTIVES

1. Obtain a greater RR to CT and PFS in patients with advanced NSCLC who receive cisplatin- and paclitaxel-based CT combined with a 45-mg/m2 daily dose of atRA with an acceptable toxicological profile .
2. Evaluate the benefit of RAR beta and RAR alfa expression as a response biomarker.

METHODS Three hundred and thirty patients with advanced NSCLC will be included to receive Paclitaxel 175 mg/m2 and Cisplatin 80 mg/m2 (PC) every 21 days for 6 cycles. Patients will be randomized to receive ATRA 45 mg2/day or placebo 1 week before treatment until completing six cycles. Imaging studies will be performed prior and after two cycles of CT to assess response. RAR beta and RAR alfa expression will be analyzed by immunohistochemistry in lung tumoral tissue and in the adjacent lung tissue.

DETAILED DESCRIPTION:
BACKGROUND Platinum-based chemotherapy (CT) is the standard treatment for advanced non-small-cell lung cancer (NSCLC). Unfortunately, the survival and response rate (RR) to CT is poor. There is great interest in new treatment strategies. One of this new strategies include the use of retinoids such as atRA. The synergistic effect of cytotoxic agents with retinoids has been demonstrated in lung cancer. At the INCan, our work group carried out a phase II study trial that included 107 patients with advanced NSCLC. They were randomized to receive atRA (20-mg/m2) or placebo combined with 80 mg/m2 of cisplatin and 175 mg/m2 of paclitaxel. The results showed a significant increase in the RR of the atRA group, reaching 55.8% ( 95% CI; 46.6-64.9%) compared with 25.4% (95% CI, 21.3-29.5%; p = 0.001) in patients who received placebo. Median Progression-free survival (PFS) in the atRA group was 8.9 months, while for those of placebo, PFS was 6.0 months (p = 0.008). There were no significant differences in the grade 3-4 side effects between groups, except for hypertriglycemia, which presented with greater frequency in the atRA group (p = 0.05). Immunohistochemical stains determine the RAR beta 2 expression in 6 of 60 tumor samples analyzed; however, all samples expressed RAR beta 2 in adjacent normal tissue.

HYPOTHESIS Patients with NSCLC who receive the scheme combined with first-line CT plus 45 mg/m2 of atRA will have a greater PFS and RR to CT with an acceptable toxicological profile.

OBJECTIVES

1. Obtain a greater RR to CT and PFS in patients with advanced NSCLC who receive cisplatin- and paclitaxel-based CT combined with a 45-mg/m2 daily dose of atRA with an acceptable toxicological profile .
2. Evaluate the benefit of RAR beta and RAR alfa expression as a response biomarker.

METHODS Three hundred and thirty patients with advanced NSCLC will be included to receive Paclitaxel 175 mg/m2 and Cisplatin 80 mg/m2 (PC) every 21 days for 6 cycles. Patients will be randomized to receive ATRA 45 mg2/day or placebo 1 week before treatment until completing six cycles. Imaging studies will be performed prior and after two cycles of CT to assess response. RAR beta and RAR alfa expression will be analyzed by immunohistochemistry in lung tumoral tissue and in the adjacent lung tissue.

POPULATON AND SAMPLE

The institutions that will recruit patients will be the National Institute of Cancerology (INCan) and the National Institute of Respiratory Diseases (INER) according to the inclusion and exclusion criteria of the protocol:

Inclusion criteria: Patients with advanced NSCLC (stages III B or IV according to the Tumor node metastasis [TNM] classification) who receive paclitaxel 175 mg/m2- and cisplatin-based palliative therapy every 3 weeks during 4 cycles; general status with a Karnofsky score of ≥70%, Eastern Cooperative Oncology Group (ECOG) ≤2, hepatic and hematic cytology tests within normal ranges, and creatinine purification >75 ml per min, who accepted to participate in the study, and who signed the letter of informed consent.

Exclusion criteria: Patients with comorbidity with another type of cancer who refuse to enter the protocol; patients who require reduction of the chemotherapy dose due to alterations in their laboratory examinations; patients with a poor general health state; absence of histological diagnosis, and previous treatment with chemotherapy.

Statistical analysis With the purpose of description, the continuous variables will be expressed as arithmetic means, medians, and Standard deviations (SDs), the variable categories as proportions and 95% confidence intervals (95% CIs). Inferential comparisons will be conducted by means of the Student t test or the Mann-Whitney U test according to data distribution (normal and non-normal, respectively) determined by the Kolmogorov-Smirnov test, for example, comparison of age means between both groups. The X2 test or the Fisher exact test will be employed to evaluate significance among categorical variables, for example, both groups (atRA vs. placebo) of ECOG higher or lower than 80, stage IIIB vs. IV, history of smoking, RAR expression, and response. Statistical significance will be determined as a p value (p <0.05) with a two-tailed test. PFS and GS times will be determined from day of initiation of chemotherapy until date of death, respectively, and will be analyzed by the Kaplan-Meier test. Comparisons between groups will be performed with the log-rank test. All variables were dichotomized analyses of the survival curves. Adjustment for potential confounders will be performed by means of Cox proportion multivariate regression analysis. The SPSS version 15 (SPSS, Inc., Chicago, IL, USA) software package will be used for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced NSCLC (stages III B or IV according to the Tumor node metastasis [TNM] classification) who receive paclitaxel 175 mg/m2- and cisplatin-based palliative therapy every 3 weeks during 4 cycles,
* General status with a Karnofsky score of ≥70%,
* Eastern Cooperative Oncology Group (ECOG) ≤ 2,
* Hepatic and hematic cytology tests within normal ranges,
* Creatinine purification > 75 ml per min,
* Those who accepted to participate in the study, and who signed the letter of informed consent.

Exclusion Criteria:

* Patients with comorbidity with another type of cancer who refuse to enter the protocol,
* Patients who require reduction of the chemotherapy dose due to alterations in their laboratory examinations,
* Patients with a poor general health state
* Absence of histological diagnosis, and
* Previous treatment with chemotherapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Obtain a greater response rate to chemotherapy, and an increase in PFS and the GS of patients with advanced-stage NSCLC who receive cisplatin- and paclitaxel-based chemotherapy and a 45-mg/m2 daily dose of atRA. | 2012

SECONDARY OUTCOMES:
Demonstrate an acceptable toxicological profile of patients with advanced NSCLC who receive chemotherapy and a daily 45-mg/m2 dose of atRA. | 2013

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medical Oncology, Instituto Nacional de Cancerología, México, State of Mexico, Mexico